CLINICAL TRIAL: NCT06891430
Title: Prognosis Analysis of Three Surgical Techniques for Arthroscopic Anterior Cruciate Ligament Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24765-4-01
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: tunnel widening; Anterior Cruciate Ligament; double-bundle reconstruction; single-bundle reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ASBR Group (Experimental): Description: Patients in this group will undergo anatomical single-bundle ACL reconstruction (ASBR). The femoral and tibial tunnels will be positioned at the center of the dense fiber area of the native ACL footprint. Graft fixation will be performed using EndoButton on the femoral side and bioabsorbable screws on the tibial side.
  Interventions: Procedure: Procedure: Anatomical Single-Bundle ACL Reconstruction
- CASBR Group (Experimental): Description: Patients in this group will undergo central axial single-bundle ACL reconstruction (CASBR). The femoral and tibial tunnels will mimic the central axis of the native ACL, spanning the dense fiber structure from anteromedial to posterolateral. Graft fixation will follow the same protocol as the ASBR group.
  Interventions: Procedure: Procedure: Central Axial Single-Bundle ACL Reconstruction
- DBR Group (Experimental): Description: Patients in this group will undergo ACL double-bundle reconstruction (DBR), with separate femoral and tibial tunnels for the anterior medial bundle (AMB) and posterior lateral bundle (PLB). Graft fixation will involve independent tensioning of AMB and PLB grafts at different knee flexion angles.
  Interventions: Procedure: Procedure: Double-Bundle ACL Reconstruction

INTERVENTIONS:
Procedure: Procedure: Anatomical Single-Bundle ACL Reconstruction — Patients undergo anatomical single-bundle ACL reconstruction with femoral and tibial tunnel drilling.
  Arms: ASBR Group
Procedure: Procedure: Central Axial Single-Bundle ACL Reconstruction — Patients undergo central axial single-bundle ACL reconstruction with optimized tunnel positioning.
  Arms: CASBR Group
Procedure: Procedure: Double-Bundle ACL Reconstruction — Patients undergo double-bundle ACL reconstruction targeting AMB and PLB footprints.
  Arms: DBR Group

SUMMARY:
This study hypothesizes that the tunnel positioning and drilling direction in two single-bundle reconstruction techniques (Anatomical Single-Bundle Reconstruction, ASBR, and Central Axial Single-Bundle Reconstruction, CASBR) influence the biomechanical environment of the graft, thereby affecting graft remodeling and maturation, ultimately impacting postoperative outcomes. Studies have shown that the graft bending angle (GBA) is a critical factor affecting graft ligamentization. ASBR, with a higher GBA, may result in poorer graft maturation, while CASBR, with a lower GBA, may provide a more favorable biomechanical environment. Additionally, graft volume has been identified as an important factor influencing postoperative graft maturation. Therefore, this study also examines the double-bundle reconstruction (DBR) technique, which has a GBA similar to CASBR.

The Impact of Three Techniques on Graft Maturation Anatomical Single-Bundle Reconstruction (ASBR)

ASBR involves drilling a single tunnel at both the femoral and tibial ends, with the tunnel positioned at the center of the dense fiber area of the ACL footprint. The femoral tunnel is positioned at 90° knee flexion and drilled at 120°, while the tibial tunnel is positioned at 70° knee flexion. Due to the higher GBA in ASBR, the graft may experience greater bending stress during motion, leading to impaired graft maturation, limited ligamentization, and increased stress concentration around the tunnel, potentially causing tunnel widening.

Central Axial Single-Bundle Reconstruction (CASBR)

CASBR also involves drilling a single tunnel at both ends, but the tunnel is positioned in the posterior region of the dense fiber area of the ACL footprint, mimicking the central axis of the native ACL. The femoral tunnel is positioned at 90° knee flexion and drilled at 120°, while the tibial tunnel is positioned at 70° knee flexion. Compared to ASBR, CASBR's lower GBA results in more uniform graft stress distribution, promoting better graft maturation and reducing the risk of stress concentration and tunnel widening.

Double-Bundle Reconstruction (DBR)

DBR involves drilling two tunnels at both the femoral and tibial ends, targeting the dense fiber areas of the anterior medial bundle (AMB) and posterior lateral bundle (PLB) of the ACL footprint. The positioning of the PLB tunnel is similar to CASBR, while the AMB tunnel is located in the anterior region of the footprint. DBR provides a more anatomically accurate distribution of forces, leading to a more even biomechanical environment. However, the increased number of tunnels may complicate stress distribution.

Impact on Postoperative Outcomes ASBR, with its higher GBA, may lead to poor graft maturation and increased tunnel widening. CASBR, with a lower GBA, offers a more favorable biomechanical environment for graft maturation. While DBR ensures a more uniform force distribution, the additional tunnels may introduce complexities in stress distribution, potentially affecting postoperative recovery and return to sports (RTS).

DETAILED DESCRIPTION:
Hypothesis and Background This study hypothesizes that the tunnel positioning and drilling direction of two single-bundle reconstruction techniques influence the biomechanical environment of the graft, which may affect graft remodeling. Poor biomechanical environments could result in suboptimal graft maturation and worse return-to-sport (RTS) outcomes. Previous research has identified the graft bending angle (GBA) as a risk factor for graft ligamentization. Anatomical Single-Bundle Reconstruction (ASBR) is associated with a higher GBA, whereas Central Axial Single-Bundle Reconstruction (CASBR) has a relatively lower GBA. Recent studies have also highlighted the influence of graft volume on postoperative graft maturation. Therefore, this section further discusses ACL double-bundle reconstruction (DBR), which has a GBA similar to CASBR. The anatomical and directional terminologies used in this study are based on the ESSKA scientific seminar on ACL reconstruction held at Imperial College London.

Techniques Anatomical Single-Bundle Reconstruction (ASBR)

ASBR involves drilling single femoral and tibial tunnels, both positioned at the center of the dense fiber area of the native ACL footprint. This technique represents the anatomical location of the ACL.

Femoral Tunnel: Positioned arthroscopically through the anteromedial portal at 90° knee flexion, targeting the center of the ACL femoral footprint. A guidewire is used without a positioning device, and the femoral tunnel is drilled at 120° knee flexion.

Tibial Tunnel: Positioned arthroscopically through the anteromedial portal at 70° knee flexion using the Smith & Nephew tibial tunnel guide. The tibial tunnel is drilled at the center of the ACL tibial footprint, with angles adjusted to 55° relative to the horizontal plane and 30° medially from the sagittal plane.

Central Axial Single-Bundle Reconstruction (CASBR)

CASBR also involves single femoral and tibial tunnels, but the tunnel positions mimic the central axis of the native ACL, spanning the dense fiber structure from anteromedial to posterolateral.

Femoral Tunnel: Positioned arthroscopically at 90° knee flexion through the anteromedial portal, targeting the posterior 60% of the ACL femoral footprint. The tunnel is drilled at 120° knee flexion.

Tibial Tunnel: Positioned arthroscopically at 70° knee flexion through the anteromedial portal using the Smith & Nephew tibial tunnel guide. The tunnel is drilled at the posterior 40% of the ACL tibial footprint, with angles adjusted to 50° relative to the sagittal plane and 40° medially from the tibial tubercle sagittal plane.

Double-Bundle Reconstruction (DBR)

DBR involves drilling two tunnels at both the femoral and tibial sides to reconstruct the anterior medial bundle (AMB) and posterior lateral bundle (PLB) of the ACL.

PLB Tunnels: The femoral tunnel is positioned at the anterior 40% of the ACL femoral footprint at 90° knee flexion and drilled at 120°. The tibial tunnel follows the CASBR tibial tunnel positioning.

AMB Tunnels: The femoral tunnel follows CASBR positioning, while the tibial tunnel is positioned at the anterior 60% of the ACL tibial footprint at 65° relative to the horizontal plane and 40° medially from the tibial tubercle sagittal plane.

Biomechanical Differences and Graft Maturation Biomechanical variations among these techniques significantly influence graft maturation and tunnel widening.

ASBR: The higher GBA results in increased bending stress on the graft, potentially impairing graft maturation and ligamentization. This stress may also lead to higher stress concentrations around the tunnel, increasing the risk of tunnel widening.

CASBR: The lower GBA provides a more favorable biomechanical environment with more uniform stress distribution. This reduces stress concentrations and minimizes the risk of tunnel widening, promoting better graft maturation.

DBR: While DBR offers a more anatomically accurate force distribution, the additional tunnels may complicate stress distribution and pose a risk of stress concentration, particularly at the bone bridges between the tunnels.

Postoperative Rehabilitation Protocol

All three surgical techniques followed the same standardized postoperative rehabilitation protocol, which has been consistently used in our institution to ensure uniformity across patient groups. The protocol includes the following components:

Knee Flexion: Patients begin knee flexion exercises on postoperative day 5, reaching 90° initially. Flexion angles are increased every two days, with a goal of 120° by six weeks and full flexion by three months.

Weight-Bearing: No weight-bearing is allowed for the first six weeks. Full weight-bearing walking is permitted after six weeks, but walking distances are minimized until three months.

Bracing: A knee brace is immediately applied postoperatively at 0° flexion. The brace is worn continuously for six weeks, except during flexion exercises. After six weeks, braces are only required outdoors, and no bracing is needed after three months.

Physical Activity: Normal walking is allowed within four months, but distances are limited. Running is restricted to 50 meters of slow jogging until six months postoperatively. High-impact sports are only permitted after nine months, provided that quadriceps strength reaches at least 80% of the contralateral side, hamstring-to-quadriceps strength ratio exceeds 85%, proprioception training is completed, and the patient undergoes sport-specific adaptation exercises for 2-3 months.

Conclusion The consistent use of this rehabilitation protocol ensures comparability across surgical techniques and minimizes variability in recovery. However, the biomechanical differences among ASBR, CASBR, and DBR highlight their distinct effects on graft maturation and tunnel widening. CASBR, with its more favorable biomechanical environment, appears to offer the best balance between graft maturation and minimal tunnel widening, while ASBR and DBR may require careful consideration of their respective biomechanical challenges.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with anterior cruciate ligament (ACL) rupture; Age between 18-50 years; All patients must have isolated anterior cruciate ligament (ACL) rupture; Knee joint degeneration < KL grade II, and intraoperative cartilage injury < ICRS grade III; All isolated ACL rupture patients must not have other ligament injuries; If accompanied by meniscus injury, the proportion of medial or lateral meniscus resection during surgery must not exceed 40%; The duration of the condition must be within one year after injury; No restriction on body weight; The cause of ACL rupture must be sports-related trauma or twisting injuries, excluding car accident injuries.

Exclusion Criteria:

Patients with other surgical contraindications; Patients with poor compliance; Patients planning pregnancy; Patients deemed unsuitable for inclusion by the researchers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
tunnel widening | From two days postoperatively to two years postoperatively
  Tunnel widening is measured as the percentage change in cross-sectional area of the graft tunnel. Using CT and MRI, we measure the cross-sectional area perpendicular to the graft tunnel two days after surgery (baseline) and again during follow-up. The tunnel enlargement rate is calculated as:
  Tunnel Enlargement Rate = (Follow-up Tunnel Area - Postoperative Day 2 Tunnel Area) / Postoperative Day 2 Tunnel Area × 100%
  The measurement unit is percentage (%), with higher percentages indicating greater tunnel widening.

SECONDARY OUTCOMES:
Return to sport | Follow-up more than two years postoperatively.
  The Return to Sport (RTS) Safety Assessment evaluates functional recovery following ACL reconstruction through comprehensive testing of muscle strength and functional performance.
  Testing includes:
  Isokinetic quadriceps strength tests at 60°/s using an electromechanical dynamometer (Biodex System III dynamometer, Biodex Medical Systems) Four types of single-legged hop tests Each participant receives a demonstration and two practice sessions prior to the formal tests, which occur 20 minutes post-exercise. All tests are performed on both the injured and uninjured legs.
  The measurement unit is the Leg Symmetry Index (LSI), calculated as a percentage (%) by comparing the performance of the injured leg to the uninjured leg. The final score is recorded as the mean LSI% across both the hop and isokinetic tests. An LSI of 100% indicates perfect symmetry between legs, with higher percentages representing better functional recovery.
IKDC 2000 | Recorded preoperatively and at follow-up more than two years postoperatively.
  The IKDC 2000 Subjective Knee Evaluation is a patient-reported outcome measure that assesses symptoms, sports activities, and function. The preoperative score is measured as baseline data for comparability, and the follow-up score after more than two years postoperatively is used to compare clinical outcomes among the three surgical techniques.
  The measurement unit is a standardized score ranging from 0 to 100, where 0 represents the lowest level of function and highest level of symptoms, and 100 represents the highest level of function and lowest level of symptoms.
Lyholm score | Recorded preoperatively and at follow-up more than two years postoperatively.
  The Lysholm Knee Scoring Scale evaluates knee function in activities of daily living. The preoperative score is measured as baseline data for comparability, and the follow-up score after more than two years postoperatively is used to compare clinical outcomes among the three surgical techniques.
  The measurement unit is a numerical score ranging from 0 to 100, where 0 represents severe knee problems and 100 represents normal knee function.
Tegner | From two days postoperatively to two years postoperatively
  The Tegner Activity Scale assesses activity level specifically related to knee function. The preoperative score is measured as baseline data for comparability, and the follow-up score after more than two years postoperatively is used to compare functional recovery among the three surgical techniques.
  The measurement unit is a numerical score ranging from 0 to 10, where 0 represents disability due to knee problems and 10 represents participation in competitive sports at a national or international elite level.

IPD SHARING:
Plan to Share IPD: Undecided
The decision not to share clinical trial results publicly is primarily driven by the need to protect patient privacy and comply with ethical and legal standards. Even with anonymization, there is a potential risk of re-identification, especially in studies involving small or unique populations. Additionally, unpublished results may involve incomplete data, ongoing analyses, or findings that require further validation to ensure accuracy and reliability. Sharing such data prematurely could lead to misinterpretation or misuse. Therefore, withholding results in certain cases is a precaution to safeguard patient confidentiality and maintain the scientific integrity of the research.